CLINICAL TRIAL: NCT04791384
Title: Multicenter Open Label Phase Ib/II Trial of Abemaciclib and Elacestrant in Patients With Brain Metastasis Due to HR+/Her2- Breast Cancer
Brief Title: Phase Ib/II Trial of Abemaciclib and Elacestrant in Patients With Brain Metastasis Due to HR+/Her2- Breast Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Criterium, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Lilly-I3Y-US-I026
Record Dates: First submitted 2020-12-30; First posted 2021-03-10 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — abemaciclib; elacestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Abemaciclib/Elacestrant (Experimental): Abemaciclib and Elacestrant combination
  Interventions: Drug: Abemaciclib; Drug: Elacestrant

INTERVENTIONS:
Drug: Abemaciclib — taken orally
  Other Names: Verzenio
Drug: Elacestrant — taken orally

SUMMARY:
This is a multi-institutional, single arm, open label, Phase Ib/II study of abemaciclib in combination with elacestrant in patients with HR+/Her2- breast cancer metastatic to the brain. Patients may have received up to two prior lines of systemic chemotherapy for locally advanced or metastatic disease. There will be no limit on prior use of endocrine therapy including aromatase inhibitors, tamoxifen and fulvestrant, given a documented clinical benefit of elacestrant in this setting.

DETAILED DESCRIPTION:
This is a multi-institutional, Phase Ib/II study in patients with HR+/Her2- breast cancer metastatic to the brain. Patients may have received up to two prior lines of systemic chemotherapy for locally advanced or metastatic disease. There will be no limit on prior use of endocrine therapy including aromatase inhibitors, tamoxifen and fulvestrant, given a documented clinical benefit of elacestrant in this setting. Single agent abemaciclib at a dose of 150 mg twice a day and elacestrant at a dose of 400mg / day will be administered to all patients, with allowances for up to 2 dose reductions due to treatment related toxicities. Patients will be evaluated for treatment emergent adverse events (AEs) during study participation, and toxicity will be assessed according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events, Version 5.0. After accrual of first 10 patients, the accrual will be halted and safety analysis (phase IB) will be performed. If response to the combination therapy will be documented in 2 or less patients accrual will be stopped. If at least 3 patients will have a documented response to therapy, accrual will continue to complete Stage 2

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible for inclusion in this study if all of the following criteria apply:

  1. Post-menopausal women with histologically or cytologically diagnosed metastatic HR+/Her2- breast cancer defined as positive for estrogen receptor or progesterone receptor (more than 1% staining by immunohistochemistry, as defined in 2010 ASCO recommendations, Hammond 2010) and negative for HER2 amplification (immunohistochemistry result of 0-1+, or a negative in situ hybridization).

     Post-menopausal status is defined as:
     1. Documented surgical bilateral oophorectomy
     2. Age > 59 years with amenorrhea for > 1 year since last menses
     3. Age < 60 years with amenorrhea for > 1 year since last menses and serum estradiol and FSH in post-menopausal laboratory range.
  2. Patients must have measurable brain metastasis (patients with leptomeningeal disease and measurable parenchymal disease are permitted) with documented intracranial disease progression. One measurable lesion >10mm, or previously irradiated lesion with increase in size by at least 5mm as defined by RANO-BM criteria and revised RECIST criteria (version 1.1, Appendix C). Patients with prior whole brain radiotherapy are permitted.
  3. Prior treatment with up to two lines of systemic chemotherapy for metastatic disease and two weeks from any previous anticancer therapy including biologics and recovered from expected toxicity; at least 4 weeks from major surgery and recovered; at least 3 weeks from radiation affecting more than 25% of bone marrow and recovered; and 2 weeks from other palliative radiation and recovered.
  4. ECOG performance status ≤ 2 (see Appendix B).
  5. Patients who received chemotherapy must have recovered (Common Terminology Criteria for Adverse Events [CTCAE] Grade ≤1) from the acute effects of chemotherapy except for residual alopecia or Grade 2 peripheral neuropathy prior to randomization. A washout period of at least 14 days is required between last chemotherapy dose and randomization (provided the patient did not receive radiotherapy
  6. Patients who received adjuvant radiotherapy must have completed and fully recovered from the acute effects of radiotherapy. A washout period of at least 14 days is required between end of radiotherapy and randomization.
  7. The patient has adequate organ function for all of the following criteria, as defined in Table 1 below.

     Table 1: Laboratory Value Guidance to Establish Adequate Organ Function System Laboratory Value Hematologic ANC: >/= 1.5 × 109/L Platelets: >/=100 × 109/L Hemoglobin: >/=8 g/dL

     Patients may receive erythrocyte transfusions to achieve this hemoglobin level at the discretion of the investigator. Initial treatment must not begin earlier than the day after the erythrocyte transfusion.

     Hepatic Total bilirubin: </= 1.5 × ULN Patients with Gilbert's syndrome with a total bilirubin </=2.0 times ULN and direct bilirubin within normal limits are permitted.

     ALT and AST: </= 3 × ULN

     Renal Serum creatinine: </= 1.5 × ULN Abbreviations: ALT = alanine aminotransferase; ANC = absolute neutrophil count; AST = aspartate aminotransferase; ULN = upper limit of normal.
  8. Ability to take oral medications.
  9. Women of child-producing potential must agree to use effective contraceptive methods prior to study entry, during study participation, and for at least 30 days after the last administration of study medication. A serum pregnancy test within 72 hours prior to the initiation of therapy will be required for women of childbearing potential.
  10. Have the ability to understand the requirements of the study, provide written informed consent which includes authorization for release of protected health information, abide by the study restrictions, and agree to return for the required assessments.
  11. Availability of archival tumor tissue (core biopsy or surgical tumor blocks) for analysis. Sites will be asked to submit archival tissue (subjects may start the study if tissue is available at an outside hospital, but not yet requested or received).

Exclusion Criteria:

* Patients will not be eligible for inclusion in this study if any of the following criteria apply:

  1. Women who are pregnant or lactating and men.
  2. Patients under age of 18
  3. Prior use of abemaciclib or elacestrant (use of other cdk4/6 inhibitors are allowed)
  4. The patient has serious preexisting medical condition(s) that would preclude participation in this study (for example, interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline Grade 2 or higher diarrhea).
  5. The patient has active bacterial infection (requiring intravenous [IV] antibiotics at time of initiating study treatment), fungal infection, or detectable viral infection (such as known human immunodeficiency virus positivity or with known active hepatitis B or C [for example, hepatitis B surface antigen positive]. Screening is not required for enrollment.
  6. The patient has a personal history of any of the following conditions: syncope of cardiovascular etiology, ventricular arrhythmia of pathological origin (including, but not limited to, ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest.
  7. Wome who are pre-menopausal (women with chemically induced menopause are eligible).
  8. More than two seizures in the last 4 weeks.
  9. Have uncontrolled serious medical or psychiatric illness.
  10. Have any medical condition that would impair the administration of oral agents including recurrent bowel obstructions, inflammatory bowel disease or uncontrolled nausea, vomiting. Baseline grade 2 or greater diarrhea.
  11. Have an additional malignancy diagnosed within 5 years of study enrollment with the exception of basal or squamous cell skin cancer or cervical cancer in situ.
  12. Patients may not be receiving any other investigational agents. A washout period of 14 days is required for all prior anti-cancer therapies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-04-21 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
The number of patients in Phase 1b part of the study with any adverse events (AE). | 1.5 years
  To determine the safety and tolerability of the abemaciclib and elacestrant combination. We will assess the incidence, nature and severity of all adverse events (AE) that occur on or after C1D1 of therapy, AE severities will be classified using the CTCAE criteria.
Assess the efficacy of the drug combination abemaciclib and elacestrant. | The whole study- 2.5 years
  Determine the overall intracranial response rate (OIRR; complete and partial response) and clinical benefit rate (CBR) as defined by brain metastasis response criteria (RANO-BM) in women with HR+ / Her2- breast cancer using the sum of study participants who experience complete response or partial response within 24 weeks or less. This assessment will look at tumor responses conducted before patients start treatment, at timepoints while receiving treatment, and at treatment end.

SECONDARY OUTCOMES:
Evaluate tumor response rates of treatment with abemaciclib and elacestrant combination. | 2.5 years
  Per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. tumor responses conducted before patients start treatment, at timepoints while they receive treatment, and when their treatment ends, will be evaluated.
Evaluate duration of tumor response rates of treatment with abemaciclib and elacestrant combination. | 2.5 years
  Duration of intracranial benefit rate will be measured per the response assessment in neuro-oncology brain metastases (RANO-BM) for the time of participation in the study.
The percentage of patients to complete the study. | 2.5 years
  Study participants will be followed for the duration of their participate in the study for overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kabos, MD, Principal Investigator — University of Colorado, Denver
Locations (3):
- United States (3):
  - University of Colorado, Aurora, Colorado
  - Duke Cancer Center, Durham, North Carolina
  - Cancer Care Northwest, Spokane Valley, Washington